CLINICAL TRIAL: NCT00252083
Title: Planned Parenthood Center of El Paso Adopting and Demonstrating the Adaptation of Prevention Techniques With Popular Opinion Leader (ADAPT-POL)
Brief Title: ADAPT-POL: Planned Parenthood Center of El Paso Adopting and Demonstrating the Adaptation of Prevention Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-U65/CCU623833; U65/CCU623833-01-1
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: Seropositive; MSM; Hispanic; Popular Opinion Leader; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Popular Opinion Leader

SUMMARY:
This study will look at the following questions:

* Was there a significant difference in HIV prevention knowledge, risk reduction attitudes, norms, intentions, self efficacy, number of sexual partners, and incidence of unprotected anal intercourse among seropositive Hispanic men who have sex with men (MSM) after the implementation of ADAPT-POL?

Hypothesis: There will be a significant increase in HIV prevention knowledge, intentions, and self efficacy concerning condom use. There will be a decrease in risk attitudes, norms, number of sexual partners, and incidence of unprotected anal intercourse among seropositive Hispanic MSM after the implementation of ADAPT-POL.

* How is exposure to the intervention and intervention dosage related to the following variables: HIV prevention knowledge, attitudes, intentions, and behaviors concerning unprotected anal intercourse?

Hypothesis: Intervention exposure and dosage are positively correlated with improved HIV prevention knowledge, attitudes, intentions, and behaviors concerning unprotected anal intercourse.

DETAILED DESCRIPTION:
The proposed project, Adopting and Demonstrating the Adaptation of Prevention Techniques (ADAPT), has two main goals: first, to assist the Centers for Disease Control and Prevention (CDC) to better understand the processes needed for adapting evidence-based behavioral interventions to fit new conditions or target populations; second, to utilize the CDC's draft adaptation guidance to adapt Jeff Kelly's Popular Opinion Leader (POL) for use with adult, seropositive Hispanic men who have sex with other men (MSM). The target population will directly participate in all phases of the intervention adaptation process.

ADAPT, known as ADAPT-POL in El Paso, will include formative research and outcome monitoring. Throughout both periods, the ADAPT-POL staff will conduct process monitoring and evaluation to assess the delivery of the intervention, and to help the CDC understand how the draft adaptation guidance procedures work in a real world setting. Representatives of the target population will participate in focus groups, key informant interviews, and community advisor meetings during the formative phase; and potentially serve as popular opinion leaders (POLs) during the implementation phase.

The knowledge obtained during the ADAPT-POL intervention will be diffused to other interventions and programs at the Planned Parenthood Center of El Paso (PPCEP). This will allow PPCEP management and staff to make informed decisions about the adoption of interventions and what steps might be necessary to adapt existing and future PPCEP interventions that target Hispanic populations. At the conclusion of ADAPT activities, the CDC-developed draft adaptation guidance will be revised based on lessons learned.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* Men who have sex with other men
* Sexual contact to orgasm with a man within past year
* Hispanic
* At least 18 years of age
* Those who frequent viable venues for recruiting pre-and post-implementation questionnaire respondents.

Exclusion Criteria:

* MSM who are not willing to identify themselves to study staff as seropositive Hispanic MSM may be excluded.
* Those under 18 years of age will be excluded from participation due to the study design precluding direct applicability of hypotheses and intervention to both adults and children due to different cognitive development, HIV prevalence levels, and social networks.
* Serious mental illness which makes the individual unsuitable for participation
* Under the influence of drugs or alcohol which makes the individual unsuitable for participation
* Anyone who does not meet the inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
reduced incidence of unprotected anal intercourse | 6 months

SECONDARY OUTCOMES:
reduced number of sexual partners engaging in unprotected anal intercourse | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vel S McKleroy, MPH, BSW, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Planned Parenthood Center of El Paso, El Paso, Texas, United States